CLINICAL TRIAL: NCT00805818
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study of NNZ-2566 in Patients With Traumatic Brain Injury
Brief Title: Study of NNZ-2566 in Patients With Traumatic Brain Injury
Acronym: INTREPID2566
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neuren Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Neu-2566-TBI-001
Record Dates: First submitted 2008-12-08; First posted 2008-12-10 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries | interventions — trofinetide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NNZ-2566 (Experimental): 20 mg/kg intravenous bolus infusion over 10 minutes followed by a continuous intravenous infusion of 1 mg/kg/h (Cohort 1, n=20), 3 mg/kg/h (Cohort 2, n=20) or 6 mg/kg/h (Cohort 3, n=133) intravenous infusion for a total of 72 consecutive hours.
  Interventions: Drug: NNZ-2566
- Sodium Chloride (0.9%) for Injection (Placebo Comparator): Intravenous bolus infusion over 10 minutes followed by a continuous intravenous infusion (Cohort 1, n=10), (Cohort 2, n=10) or (Cohort 3, n=67) intravenous infusion for a total of 72 consecutive hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NNZ-2566 — Solution for intravenous infusion.
  20 mg/kg intravenous bolus infusion over 10 minutes followed by a continuous intravenous infusion of 1, 3, or 6 mg/kg/h for a total of 72 consecutive hours.
  Other Names: Glycyl-L-2-Methylprolyl-L-Glutamic Acid
  Arms: NNZ-2566
Drug: Placebo — Sodium Chloride 0.9% Injection
  Other Names: Sodium Chloride 0.9% Injection
  Arms: Sodium Chloride (0.9%) for Injection

SUMMARY:
The purpose of this study is to determine whether NNZ-2566 is safe and effective in the treatment of Traumatic Brain Injury (TBI).

DETAILED DESCRIPTION:
Moderate to severe traumatic brain injury frequently results in persistent problems with memory, attention span, mood and more complex brain functioning such as planning and organizing. There are currently no drugs available to reduce the brain damage or the persisting symptoms that result from TBI. The longer term goal of this study is to provide physicians with a safe and effective treatment for TBI.

ELIGIBILITY:
Inclusion Criteria:

* Non-penetrating TBI.
* Male.
* Age 18-70 years.
* Admission to hospital.
* Post resuscitation GCS 4-12.
* Have at least one reactive pupil.
* Randomization within 7 hours of injury with the ability to receive investigational product within 8 hours of injury.
* Hemodynamically stable after resuscitation (systolic blood pressure (SBP) >100 mm Hg).
* Willing to undergo all neuropsychological and activities of daily living (ADL) testing (i.e. understand English, able to read, write, have sufficient motor dexterity and, be available for follow-up visits at 4-6 weeks and 12-14 weeks post injury).

Exclusion Criteria:

* Penetrating brain injury.
* Spinal cord injury.
* Presence or known history of prior cerebral injury requiring hospitalization that would, in the opinion of the Investigator, interfere with or bias the assessment of efficacy.
* Non-traumatic brain injury.
* Known history of any medical or psychiatric disorder, or any severe concomitant disease, that in the opinion of the Investigator would interfere with or bias the assessment of efficacy. This includes the following: schizophrenia; bipolar disorder; major depressive disorder; post traumatic stress disorder (PTSD); generalized anxiety disorder; attention deficit hyperactivity disorder; neurodegenerative diseases (Alzheimer's, Parkinson's, Huntington's disease, vascular dementia, Diffuse Lewy Body Disease); stroke; brain tumor; multiple sclerosis (MS); seizure disorders; chronic pain disorder; alcoholism or substance abuse.
* Significant non-central nervous system (CNS) injuries sustained at the time of the TBI that in the opinion of the Investigator would interfere with or bias the assessment of efficacy.
* Weight >150 kg.
* Participation in another clinical trial within the previous 4 weeks.
* Clinical state requiring greater than 6 L colloid or crystalloid fluid resuscitation prior to randomization.
* Inability to obtain informed consent from legally acceptable representative.
* Prior enrollment in this study.
* QTc Exclusions. The study will use the exclusion criteria as defined in ICH Guideline E14 to exclude patients with a risk of QT/QTc prolongation, as follows:

  * A marked baseline prolongation of corrected QT/QTc interval >450 ms.
  * History of risk factors for torsade de pointes (e.g. heart failure, hypokalemia (serum potassium at screening (<3.0 mmol/L)or family history of long QT syndrome).

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2010-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Reduced incidence, compared to placebo, of adverse events (AEs) and serious adverse events (SAEs) | AEs to discharged or Day 30 post randomization, whichever occurs first, and SAEs through to 3 months (defined as 12-14 weeks), post randomization.

SECONDARY OUTCOMES:
Evidence of efficacy in modifying global outcomes by evaluating Glasgow Outcome Scale - Extended (GOS-E) and activities of daily living (Mayo-Portland Adaptability Inventory - 4th Edition (MPAI-4)) | 1 month (defined as 4-6 weeks) and 3 months (defined as 12-14 weeks), post randomization.
Improvement in cognitive and neuropsychological functioning. | 1 month (defined as 4-6 weeks) and at 3 months (defined as 12-14 weeks), post randomization.
Modification of the acute physiological processes in TBI by evaluating electroencephalographic (EEG) determinants in patients with moderate to severe TBI (defined as GCS 4-12), and biomarker levels. | Baseline through to 72 hours post-start of infusion.
Blood pharmacokinetics (PK) of an intravenous (i.v) dose of NNZ-2566 when administered as a 10-minute infusion immediately followed by a 72-hour infusion. | Start of infusion through to 12 hours post infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Ross R Bullock, M.D., PhD, Principal Investigator — University of Miami, Lois Pope Life Center
Locations (20):
- United States (20):
  - University of South Alabama, Mobile, Alabama
  - University of Arizona, Tucson, Arizona
  - Arrowhead Regional Medical Center, Colton, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - University of California, Davis Medical Center, Sacramento, California
  - University of Miami, Lois Pope Life Center, Miami, Florida
  - The Queen's Medical Center, Honolulu, Hawaii
  - Our Lady of the Lake Hospital, Baton Rouge, Louisiana
  - Detroit Receiving Hospital and University Health Center, Detroit, Michigan
  - Sinai Grace Hospital, Detroit, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - SUNY Upstate Medical University, Syracuse, New York
  - University of Cincinnati, Mayfield Clinic, Cincinnati, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - St Luke's University Hospital, Bethlehem, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Texas Health Harris Methodist Hospital Fort Worth, Fort Worth, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Charleston Area Medical Center, Charleston, West Virginia
  - University of Wisconsin, Froedtert Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee JW. The EEG Ictal-Interictal Continuum-A Metabolic Roar But a Whimper of a Functional Outcome. Epilepsy Curr. 2019 Jul-Aug;19(4):234-236. doi: 10.1177/1535759719855968. Epub 2019 Jun 14. PMID 31198061
- [Derived] Lee H, Mizrahi MA, Hartings JA, Sharma S, Pahren L, Ngwenya LB, Moseley BD, Privitera M, Tortella FC, Foreman B. Continuous Electroencephalography After Moderate to Severe Traumatic Brain Injury. Crit Care Med. 2019 Apr;47(4):574-582. doi: 10.1097/CCM.0000000000003639. PMID 30624278
- See also: Click here for more information about this study — http://www.neurenpharma.com